CLINICAL TRIAL: NCT03983811
Title: Adjuvant Chemotherapy of EGFR-Mutated Non-Small Cell Lung Cancer Patients With or Without Intercalated Icotinib Therapy: a Randomized, Placebo-controlled Trial
Brief Title: Adjuvant Chemotherapy With or Without Intercalated Icotinib
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Kaican Cai, Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NFEC-2019-077
Record Dates: First submitted 2019-06-09; First posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — icotinib; Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy+Icotinib (Experimental): Patients receive 4 cycles of platinum-based doublet chemotherapy on day 1 with intercalated icotinib (D8-15) every 3 weeks, and continued icotinib for 2 years or until the occurrence of disease relapse, metastasis or unacceptable icotinib or chemotherapy toxicity
  Interventions: Drug: Icotinib; Other: chemotherapy
- Chemotherapy+Placebo (Placebo Comparator): Patients receive 4 cycles of platinum-based doublet chemotherapy on day 1 with intercalated placebo (D8-15) every 3 weeks, and continued placebo for 2 years or until the occurrence of disease relapse, metastasis or unacceptable toxicity
  Interventions: Drug: Placebo; Other: chemotherapy

INTERVENTIONS:
Drug: Icotinib — Patients receive 4 cycles of platinum-based doublet chemotherapy on day 1 with intercalated icotinib (D8-15) every 3 weeks, and continued icotinib for 2 years or until the occurrence of disease relapse, metastasis or unacceptable icotinib or chemotherapy toxicity
  Arms: Chemotherapy+Icotinib
Drug: Placebo — Patients receive 4 cycles of platinum-based doublet chemotherapy on day 1 with intercalated placebo (D8-15) every 3 weeks, and continued placebo for 2 years or until the occurrence of disease relapse, metastasis or unacceptable toxicity
  Arms: Chemotherapy+Placebo
Other: chemotherapy — Patients in each groups need to receive 4 cycles of platinum-based doublet chemotherapy

SUMMARY:
Epidermal growth factor receptor (EGFR) mutations occur in up to 50% of Asian patients with non-small cell lung cancer (NSCLC). Treatment of advanced NSCLC patients with EGFR-tyrosine kinase inhibitors (EGFR-TKI) confers a significant survival benefit. This study aims to assess the efficacy and safety of adjuvant chemotherapy with or without Intercalated combination of icotinib in patients undergoing resection of stage IIB to IIIA (N1-2) EGFR-mutated NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing completely resection of EGRF mutation-positive NSCLC Staging IIB to ⅢA, N1-2; PS = 0 or 1; Adequate hematological, biochemical and organ functions

Exclusion Criteria:

* Systemic anticancer therapy prior to surgery, other malignancies before or during the study, any unstable illness, women who were pregnant or lactating

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | From the date of surgery until the date of first confirmed disease relapse or metastasis, whichever came first, assessed up to 5 years
  The amount of time that patient lives without known recurrence

SECONDARY OUTCOMES:
Number of Participants with Adverse Effects | Duration of receiving chemotherapy and oral icotinib, expected to be 2.5 years